CLINICAL TRIAL: NCT01200927
Title: Investigation of the Dynamics of Sitting Postural Control in Infants With Cerebral Palsy
Brief Title: Sitting Postural Control in Infants With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0183-02-FB; H133G040118 (Other Grant/Funding Number: Dept of Education, NIDRR)
Record Dates: First submitted 2010-09-10; First posted 2010-09-14 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Palsy
Keywords: infant; sitting; postural control
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Typically Developing Infants (No Intervention): Typically developing infants (5 months old, SD .5 months at entry) were followed longitudinally as a comparison for postural variables. The primary outcome measure is Center of Pressure (COP) data, from which linear and nonlinear variables were extracted. The Gross Motor Function Measure (GMFM) sitting subsection was our clinical outcome measure.
- Home Program (Active Comparator): Home program (1x/week for 8 weeks). The primary outcome measure is Center of Pressure (COP) data, from which linear and nonlinear variables were extracted. The Gross Motor Function Measure (GMFM) sitting subsection was our clinical outcome measure.
  Interventions: Other: Physical therapy
- Perceptual-motor intervention (Active Comparator): Perceptual-motor intervention (2x/week for 8 weeks. The primary outcome measure is Center of Pressure (COP) data, from which linear and nonlinear variables were extracted. The Gross Motor Function Measure (GMFM) sitting subsection was our clinical outcome measure.
  Interventions: Other: Physical therapy

INTERVENTIONS:
Other: Physical therapy — Perceptual motor therapy, comparing twice weekly to once weekly home program
  Arms: Home Program; Perceptual-motor intervention

SUMMARY:
The overall goal of this research is to understand the mechanisms underlying the development of postural control in sitting using new methodology, in order to provide a scientific basis for evaluation and treatment of posture and movement disorders in infants with cerebral palsy. The development of early posture control remains poorly understood despite considerable therapeutic effort. Infants with cerebral palsy show their first delays in the acquisition of sitting, with subsequent problems developing adequate posture and movement control. Identifying the delay, determining the nature of the problem, and evaluating the effectiveness of treatment quickly, are vital in the early part of an infant's life, since this is the time of greatest plasticity. Tools from nonlinear dynamics, which are increasingly being used to examine other biological rhythms, are used in this study to analyze postural sway from center of pressure data during the development of sitting postural control.

DETAILED DESCRIPTION:
Background: The ability to sit independently is fundamental for function but delayed in infants with cerebral palsy (CP). Studies of intervention directed specifically toward sitting in infants with CP have not been reported. Objective: Our purpose was to compare two interventions for improving sitting postural control in infants with CP. Design: For this randomized longitudinal study, infants under 2 years old and at risk for CP were recruited for intervention directed toward sitting independence. Setting: The intervention was conducted at home or at an outpatient facility. Patients: Fifteen typically developing infants (5 months old, SD .5 months at entry) were followed longitudinally as a comparison for postural variables. Thirty-five infants with delays in achieving sitting were recruited. Infants with delays were randomly assigned to a home program (1x/week for 8 weeks; mean age=15.5 months, SD=7 months), or a perceptual-motor intervention (2x/week for 8 weeks; mean age=14.3 months, SD=3 months). Measurements: The primary outcome measure was Center of Pressure (COP) data, from which linear and nonlinear variables were extracted. The Gross Motor Function Measure (GMFM) sitting subsection was our clinical outcome measure. Results: There was a main effect of time in the GMFM sitting subscale and in two of the COP variables. Interaction of group by time factors indicated significant differences between intervention groups on two COP measures, in favor of the group with perceptual-motor intervention. Limitations: The small number of infants limits the ability to generalize the findings. Conclusions: Although both groups made progress in the GMFM, the COP measures indicated an advantage for the group with perceptual-motor intervention. The COP measures appear sensitive for assessment of infant posture control and quantifying intervention response.

ELIGIBILITY:
Inclusion Criteria:

* able to prop sit for 10 seconds
* 1.5 SD below mean on Peabody motor assessment
* between 5 months and 24 months old
* diagnosis of CP or at risk for CP

Exclusion Criteria:

* blindness
* dislocated hip

Ages: 5 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2004-12-01 (Actual); Primary Completion 2008-06-01 (Actual); Study Completion 2008-06-01 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure, Sitting Section | 2 months
  sitting skill assessment

SECONDARY OUTCOMES:
Center of pressure measures | 2 months
  linear and nonlinear measures of center of pressure in sitting

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Stergiou, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Harbourne RT, Willett S, Kyvelidou A, Deffeyes J, Stergiou N. A comparison of interventions for children with cerebral palsy to improve sitting postural control: a clinical trial. Phys Ther. 2010 Dec;90(12):1881-98. doi: 10.2522/ptj.2010132. Epub 2010 Oct 21. PMID 20966212